CLINICAL TRIAL: NCT01975714
Title: Intraocular Pressure and Tolerability Study of Preservative Free Bimatoprost 0.03% Unit Dose (BUDPF) or Preservative Free Latanoprost 0.005% Unit Dose (LUDPF) (Monoprost®) in Patients With Ocular Hypertension or Glaucoma: A Randomized, Single Masked, 3 Month Cross-over, Investigator Led, European Multicentre Trial (SPORT)
Brief Title: Intraocular Pressure and Tolerability Study of Preservative-free Prostaglandins (Bimatoprost and Latanoprost) on Glaucoma and Ocular Hypertension: European, Multicentric, Investigator-led, Single Masked Study
Acronym: SPORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Collaborators: European Vision Institute Clinical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ECR-GLC-2013-06
Record Dates: First submitted 2013-10-23; First posted 2013-11-05 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular hypertension; Preservative-free prostaglandins
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Latanoprost (Period I) + Bimatoprost (Period II) (Experimental): Preservative-free latanoprost 0.005% Unit Dose (LUDPF) (Monoprost) eye drops will be administered every day at 21:00 for the first 3 months.
  After the follow-up visit, patient will start Preservative-free bimatoprost 0.03% Unit Dose (BUDPF) eye drops every day at 21:00 for the last 3 months.
  Interventions: Drug: Preservative-free latanoprost; Drug: Preservative-free bimatoprost
- Bimatoprost (Period I) and Latanoprost (Period II) (Experimental): Preservative-free bimatoprost 0.03% Unit Dose (LUDPF) (Monoprost) eye drops will be administered every day at 21:00 for the first 3 months.
  After the follow-up visit, patient will start Preservative-free latanoprost 0.005% Unit Dose (BUDPF) eye drops every day at 21:00 for the last 3 months.
  Interventions: Drug: Preservative-free latanoprost; Drug: Preservative-free bimatoprost

INTERVENTIONS:
Drug: Preservative-free latanoprost
  Other Names: Monoprost
Drug: Preservative-free bimatoprost

SUMMARY:
Bimatoprost 0.03% preservative free monodose eye drops solution (BUDPF) is a new product composed of a synthetic prostamide, bimatoprost 0.3% in a preservative free formulation. This new product is used as a once-daily topical ocular therapy for the reduction of elevated intraocular pressure (IOP) in patients with open-angle glaucoma, or ocular hypertension, and that are sensitive to preservatives. The individual active component of BUDPF, bimatoprost is an established therapeutic agent with well documented IOP efficacy (1). Prostamides, such as bimatoprost, are believed to lower IOP mainly by increasing uveoscleral outflow. The comparator, Preservative Free Latanoprost 0.005% Unit Dose (LUDPF, eg. Monoprost®), was recently launched in a number of countries in Europe and contains latanoprost in a new preservative free formulation.

It is clinically important to compare these newly entered preservative free products with respect to tolerability and efficacy. A better tolerability combined with maximum efficacy will reduce the burden of daily glaucoma therapy and provide a clear therapeutic benefit to the glaucoma patient by providing enhanced compliance and real-world IOP-lowering efficacy.

The hypothesis of the study is that monodose bimatoprost is more effective than monodose latanoprost by at least 1 mmHg.

(AIBILI applied for an unrestricted grant from Allergan to perform this study)

ELIGIBILITY:
Inclusion Criteria includes:

* Ocular hypertension, pseudoexfoliation glaucoma (XFG) or primary open-angle glaucoma (POAG) patients that have been on a preserved prostaglandin monotherapy for at least 6 weeks. At prescreening and screening visit the IOP is less than or equal to 21 mm Hg in both eyes.

Exclusion Criteria includes:

* Any ocular condition that are of safety concern, visual field defects with an MD value above -12dB, a closed/barely open anterior chamber angles or history of acute angle closure on either eye, ocular surgery within the past three months on either eye; glaucoma surgery within the past 6 months on either eye, ocular inflammation/infection occurring within three months prior to pretrial visit on either eye, pigmentary glaucoma or neovascular glaucoma on either eye, topical ocular medication that can interfere with study medication on either eye and known hypersensitivity to any component of the trial drug solutions and participation in any other clinical trial, involving an investigational drug within one month prior to pretrial visit

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Difference in mean IOP values between the 2 groups at 6 months | 6 months

SECONDARY OUTCOMES:
Difference in IOP values IOP values, visual acuity, hyperaemia, visual acuity and tolerability between the groups in change from baseline | Month 3; Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, MD, Principal Investigator — UZ Leuven
Locations (7):
- Vienna, Austria
- Leuven, Belgium
- Italy (2):
  - Milan
  - Rome
- Coimbra, Portugal
- Geneva, Switzerland
- London, United Kingdom